CLINICAL TRIAL: NCT04244968
Title: A Study to Measure the Patient Satisfaction, Quality of Life, Health Status and Clinic Outcomes for Patients Attending MSK Triage Clinics in Rheumatology
Brief Title: Satisfaction, QoL,Health Status & Clinic Outcomes for Patients Attending MSK Triage Clinics in Rheumatology
Status: Active, not recruiting | Type: Observational
Sponsor: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Michelle Heraughty, Clinical Specialist Physiotherapist, Health Service Executive, Ireland
Other Study IDs: REC SUH 763
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Pain; Rheumatologic Disorder
Keywords: Physiotherapy Triage; Musculoskeletal Pain; Patient Satisfaction VSQ 9; MSK HQ
MeSH Terms: conditions — Musculoskeletal Pain; Collagen Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to measure the impact of musculoskeletal (MSK) complaints on the quality of life and general health of MSK Patients attending MSK triage clinics. The investigators will also record the proposed management options for patients' complaints. This will be achieved by asking patients to complete questionnaires (MSK HQ) at musculoskeletal triage clinic appointment, by undertaking a clinical assessment, by recording the proposed management plan and assessing if patients have follow up appointments for the same complaint in the following year. The investigators will also measure patient satisfaction using VSQ 9 Questionnaire. After a year the investigators will repeat the MSK HQ to assess the longterm impact of MSK Triage appointment on the MSK complaint.

DETAILED DESCRIPTION:
At present there is no data available to describe the impact of musculoskeletal (MSK) disease on the Quality of life and General Health for patients attending Rheumatology MSK triage clinics in SUH and OHLM or in similar service around Ireland. A new questionnaire (MSK HQ) has been developed which has been validated in use with this population. This will be completed by the patient on the day of the appointment and again a year later. Their number of visits to secondary care in the year after their visit will also be captured and analysed. This information will inform the health service of the outcomes of these patients and the impact of their MSK disease on the health service. It will also help with resource allocation and planning for future services, which will ensure the best service for these patients in the future.

Alongside this, Patient satisfaction and feedback is vital to ensuring service quality and quality improvement. The VSQ 9 will be used to measure Patient Satisfaction in this study to evaluate if patients are satisfied with the service they have received on the day. The repeated MSK HQ will help identify if their triage clinic appointment was beneficial to their Quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Patients who attend the musculoskeletal Triage Clinic in Rheumatology.
* Patients who can answer the study questionnaires independently.

Exclusion Criteria:

* Under 18 years
* Patients who present with red flag conditions, inflammatory disease or non-musculoskeletal conditions.
* Patients who cannot answer the study questionnaires independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending MSK Triage clinics in Rheumatology who meet the inclusion criteria outlined
Sampling Method: Non-Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal Health Questionnaire | Baseline
  Self Reported Questionnaire measuring patients health status, Score range 0 -56, with better score indicating better health status

SECONDARY OUTCOMES:
Visit-Specific Satisfaction Questionnaire version 9 | Baseline
  Patient Satisfaction Questionnaire, Score range 9 - 45, with higher scores indicating lower patient satisifaction
Change in Musculoskeletal Health Questionnaire | One year post baseline
  Self Reported Questionnaire measuring patients health status, Score range 0 -56, with better score indicating better health status

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Heraughty, MSc, Principal Investigator — HSE Ireland
Locations (1):
- Sligo University Hospital, Sligo, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill JC, Kang S, Benedetto E, Myers H, Blackburn S, Smith S, Dunn KM, Hay E, Rees J, Beard D, Glyn-Jones S, Barker K, Ellis B, Fitzpatrick R, Price A. Development and initial cohort validation of the Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) for use across musculoskeletal care pathways. BMJ Open. 2016 Aug 5;6(8):e012331. doi: 10.1136/bmjopen-2016-012331. PMID 27496243
- [Background] Kennedy DM, Robarts S, Woodhouse L. Patients are satisfied with advanced practice physiotherapists in a role traditionally performed by orthopaedic surgeons. Physiother Can. 2010 Fall;62(4):298-305. doi: 10.3138/physio.62.4.298. Epub 2010 Oct 18. PMID 21886368
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221